CLINICAL TRIAL: NCT01869140
Title: the Hypoalgesic Effect of Spinal Manual Therapy on an Healthy Population: a Randomized Clinical Trial
Brief Title: the Hypoalgesic Effect of Spinal Manual Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Franco Europeen de Chiropratique (Other)
Responsible Party: Principal Investigator, Audo, PhD stud, Institut Franco Europeen de Chiropratique
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: IFEC-001
Record Dates: First submitted 2013-05-17; First posted 2013-06-05 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Activator Appliances

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sham spinal manual therapy (Sham Comparator): activator set to zero
  Interventions: Device: spinal manual therapy
- percussive spinal manual therapy (Experimental): activator set to the maximum force
  Interventions: Device: spinal manual therapy
- Firm thoracic spinal manual therapy (Experimental): Firm thoracic manipulation
  Interventions: Device: spinal manual therapy

INTERVENTIONS:
Device: spinal manual therapy — spinal manipulation either manual or instrumental (activator)
  Other Names: activator

SUMMARY:
To study the immediate effect of spinal manual therapy on pain perception in normal subjects

DETAILED DESCRIPTION:
Is this effect only local or is it also noticed away from the stimulated area? How long does it last? Is there a dose/response phenomenon?

ELIGIBILITY:
Inclusion Criteria:

Healthy Students who volunteer from Murdoch University

-

Exclusion Criteria:

* contraindication to spinal manual therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
the Pressure pain threshold in KPa/Cm2 will be measure with an Algometer (SOMEDIC) | the pressure pain threshold will be measure immediately after intervention and every 15 minutes during 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: yannick audo, PhD student, Principal Investigator — Institut Franco Europeen de Chiropratique
Locations (1):
- Murdoch University, Perth, Western Australia, Australia